CLINICAL TRIAL: NCT02629770
Title: Clindamycin-Rifampin Interactions: Effect of Rifampin's Enzyme-induction (Cytochrome P450 3A4/3A5) on Plasma Clindamycin Concentrations, With Clindamycin Given Intravenously and Orally to Treat Bone-and-joint Infections
Brief Title: Clindamycin-rifampin Drug Interaction in the Treatment of Bone and Joint Infections
Acronym: CLIRIFA
Status: Completed | Type: Observational
Sponsor: Groupe Hospitalier Diaconesses Croix Saint-Simon (Other)
Collaborators: Fondation Ophtalmologique Adolphe de Rothschild (Network)
Responsible Party: Sponsor
Other Study IDs: VZR_2014-3
Record Dates: First submitted 2015-12-10; First posted 2015-12-14 (Estimated); Last update posted 2021-02-11 (Actual); Status verified 2021-02

CONDITIONS: Arthritis, Infectious; Bone Diseases, Infectious
MeSH Terms: conditions — Arthritis, Infectious; Bone Diseases, Infectious

STUDY DESIGN:
Observational Model: Ecologic or Community | Time Perspective: Cross-Sectional

INTERVENTIONS:
Drug: usual antibiotic treatment — pharmacological studies in patients treated with usual antibiotics, for different types of joint and bone infections

SUMMARY:
Treatment of bone and joint infections remains difficult and variable according to centres and countries. Clindamycin given intravenously and followed by an oral route is recommended for the treatment of staphylococcal, streptococcal and anaerobes bone and joint infections by the French Society for Infectious Diseases. For staphylococcal bone and implant infections, rifampin is a major drug, as it remains active in bacterial biofilm and on quiescent staphylococci. For that reasons, clindamycin-rifampin combination therapy is frequently used in these infections.Clindamycin is metabolized by the P450 3A4 cytochrome, an enzyme strongly inducible by rifampin. A retrospective study published in 2010 on 70 patients treated for bone and joint infections showed that clindamycin serum concentrations were significantly lower when clindamycin was combined with rifampin (5.3 mg/liter vs 8.9 mg/liter; p<0.02). This drug interaction could even be stronger with the oral route, because of hepatic first-past effect, ending up with very low clindamycin serum concentration, a risk of selecting resistant microorganisms and treatment failure. This latter point is an important issue, because clindamycin has an excellent oral bioavailability and is frequently used in oral regimens. In the above study, a wide variability of clindamycin serum concentration was observed in the group of patients treated with combination therapy (1-12mg/l) suggesting interindividual variability. Rifampin induction of CYP 450 3A4/A5 depends on different receptor (PXR, RXR, LXRalpha) submitted to genetic polymorphism. Hypothesis: Plasma clearance of clindamycin (CLclin) combined with rifampicin (CLclinrif) is higher when clindamycin is administered by the oral route (CLclinrif OR) compared with IV administration (CLclinrif IV).

ELIGIBILITY:
Inclusion Criteria:

* age ≥18 years
* surgical management of OAI
* Postoperative IV antibiotic therapy for 10±2 days
* Chronic bone and/or joint infection (evolving for >4 weeks) with bacteriologically documented staphylococci, streptococci or susceptible anaerobes in skin flora susceptible to clindamycin and rifampin
* Continuation of IV administration possible for a maximum of 25 days
* Patient consent to participate in the study
* Patients entitled enrolled to a French National Health Insurance

Exclusion Criteria:

* Allergy or intolerance to the family of antibiotics used, i.e. lincosamides (clindamycin, lincomycin) and rifamycins (rifampin), or to one of their constituents
* Taking active products able to induce CYP3A4/3A5: alcohol (chronic intake), anti-seizure drugs (carbamazepine, phenobarbital, phenytoin), anti-infectious agents (rifabutin, efavirenz, nevirapine, griseofulvin), anti-fungals (ketoconazole, itraconazole, voriconazole, posaconazole, fluconazole, miconazole), calcium channel blockers (diltiazem, verapamil), macrolides (erythromycin, clarithromycin, josamycin, telithromycin)
* Being treated with one of the following: cyclosporine and/or tacrolimus (immunosuppressants) ; midazolam (psychotropic agents)
* Human immunodeficiency virus-positive patient being treated with protease inhibitors (ritonavir, amprenavir, atazanavir, indinavir, nelfinavir, lopinavir, saquinavir) or delavirdine
* Cirrhosis, hepatocellular insufficiency
* Creatinine clearance < 30 mL/min (according to the cockcroft and gault formula)
* Severe sepsis (systolic blood pressure (SBP) <90 mm Hg; O2 saturation <90%, encephalopathy, oligo-anuria, creatininemia >176 mmol/L, platelets <100,000/mm3, INR >1.5, Glasgow coma score <13) or septic shock (persistent hypotension despite volumetric filling) at arrival in the unit
* Porphyria
* Congenital galactosemia, glucose and galactose malabsorption syndrome, lactase deficit because of the presence of lactose in the dalacin® capsules
* Intolerance of fructose, glucose and galactose malabsorption syndrome, sucrase-isomaltase deficit because of the presence of saccharose in the rifadin® capsules
* Major cognitive disorders, according to the DSM IV-TR (Diagnostic and Statistical Manual of Mental Disorders) definition (36)
* Weight >100 kg or <50 kg
* Woman of childbearing age using estrogen-progestin contraception and not wanting to switch to an effective mechanical-type contraceptive method
* Pregnancy or breast-feeding
* Patient under guardianship

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: patients hospitalized for medical-surgical management of OAIs in the Department of Trauma and Bone Surgery
Sampling Method: Non-Probability Sample
Enrollment: 49 (Actual)
Dates: Start 2015-12 (Actual); Primary Completion 2019-12 (Actual); Study Completion 2019-12 (Actual)

PRIMARY OUTCOMES:
mean clearances of clindamycin | 3 weeks
  The principal evaluation criterion is the mean clearances of clindamycin with and without administration of rifampin (intravenous or oral administration)
mean clearances of clindamycin | 5 weeks
  The principal evaluation criterion is the mean clearances of clindamycin with and without administration of rifampin (intravenous or oral administration)

SECONDARY OUTCOMES:
plasma concentrations of IV- or PO-administered clindamycin, combined or not with rifampin. | 3 weeks
plasma concentrations of IV- or PO-administered clindamycin, combined or not | 5 weeks

CONTACTS AND LOCATIONS:
Locations (1):
- GH Diaconesses Croix Saint Simon, Paris, Île-de-France Region, France